CLINICAL TRIAL: NCT03105635
Title: ARC - Access to Resources in the Community/Acces Aux Ressources Communautaires
Brief Title: ARC -Access to Resources in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 20160914-01H
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Problems With Access to Health Care
Keywords: Community Resources; Health Navigator

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants are patients Care providers are practices
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Participating primary care providers will be encouraged to refer their patients who could benefit from community resources to these services. They will complete the study referral form for all patients referred to a resource. They will briefly mention the study to patients who are referred to a community resource, and ask for their verbal consent to be contacted by a member of the research team to learn more about the study, and leave a "patient recruitment package" with them.
  Interventions: Other: Mixed method feasibility study
- Practice and Provider (Other): Four to six practices will be recruited to participate in this feasibility study. Primary care members working in a participating practice will be invited to participate in the study.
  All primary care providers will be encouraged to participate and at least one primary care provider is required to participate to include the practice in the study.
  After the obtaining an interest from a practice member to whom the invitation email was sent, we will offer all practice members eligible for the study an information session during which the study is described and participation offered. The practice manager or lead will be provided with the Practice Information and Consent Form
  Interventions: Other: Mixed method feasibility study

INTERVENTIONS:
Other: Mixed method feasibility study — Participating practices will receive the following:
  1. Training on community resources : An orientation regarding the availability of the local community health and social resources, and the existing navigation services that can support individuals identify the appropriate resource.
  2. Facilitation to enhance referrals: help support practices to make the desired adaptations to enhance referrals
  3. Promotional material to engagement patients: Practices will provide an area in the waiting room where promotional material on the benefit and availability of community resources will be displayed.
  4. Navigator: The services of a Navigator

SUMMARY:
Some people living with health problems require extra support to properly manage their conditions, as family doctors are only able to spend limited time in the office with these patients. There are many resources and programs in the community that can provide the necessary time and support for these patients, yet many patients are unaware that such resources exist. Patient navigators have been shown to be useful in helping patients with certain conditions (such as cancer) to get to the resources they need, especially when they have social challenges that make it difficult for them to reach these programs (for example, language or transportation barriers, poverty, or poor social support). This study will look at how helpful Navigators are to link patients at family doctors' offices to community resources. To do this, family doctors' offices in Ottawa will be recruited. All offices will receive training on referring patients to community resources, and half of these (intervention) will have a Navigator assigned to the practice. This study will assess whether access to a Navigator increases patients' access to community social and health services. In addition, the study aims to understand whether English and French speaking individuals are as likely to benefit from a Navigator in accessing community health and social services in the language of their choice.

DETAILED DESCRIPTION:
This project brings together two funding partners. The first, the Canadian Institutes of Health Research's Community Based Primary Health Care Team Grant SPOR initiative funded a five-year program of research (known as IMPACT: Innovative Models Promoting Access-to-Care Transformation, http://www.impactresearchprogram.com/). The goal of the IMPACT Project is to increase access to community-based primary health care for vulnerable populations. The lead for the Ontario arm of the IMPACT project, Simone Dahrouge, has undertaken a community engagement initiative within the Champlain Local Health Integration Network (LHIN) to understand the barriers patients face to adequately access community based resources and how these can be overcome.

The second funding partner is the Ontario Ministry of Health and Long Term Care, through the Ontario SPOR Support Unit, in support of the Working Group on Ontario's Francophone Communities. This funding support aims specifically at addressing the access needs for Ontario Francophones living in minority situations.

These two initiatives now form the Access to Resources in the Community/Accès aux Resources Communautaires (ARC) project. ARC builds upon previous activities of the IMPACT project, under the OHSN Research Ethics Board Protocol #20140131-01H and Bruyère Continuing Care Research Ethics Board Protocol #M16-14-021. That phase of the IMPACT project enabled Dr. Dahrouge and her team to develop a Local Innovation Partnership (LIP) within the Champlain LHIN. This partnership led to the assembly of a LIP Core Team in July 2015, and includes patients of various minority communities who contribute their experience and expectations, primary care providers from different care models and leaders from organizations responsible for community services (Community Care Access Centres and Community Health Centres) who inform the best approach to the integration of the two sectors, and health planners (the LHIN Primary Care Lead, senior integration specialist and others) who bring their broader context health services knowledge as well as resources (such as practice transformation facilitation services) to the project. These stakeholders have identified poor access to community based services as a priority access gap, and have selected linkage/collaboration between primary care and community resources to address this gap. The LIP Core Team is comprised of the research team, and representatives from the regional health authority (Champlain LHIN), home and community care services (Champlain Community Care Access Centre), Ontario 211, Champlain Healthline, the University of Ottawa Office of Social Accountability, local Community Health Centres, primary care providers, and community members (Additional information: 5 Champlain LIP Core Team).

The research team has also conducted several interviews and focus groups (as part of the IMPACT project) with community stakeholders to inform the approach to the ARC intervention so that it is acceptable to all. Two realist reviews have been commissioned and completed by a team of experts to help us understand the critical success factors and shape our intervention. One review is focused on "community navigators" and the other on "primary care referral to community services" to help the team understand the factors that support us. This information was used to develop the ARC intervention. A number of themes identified in these reviews including training for clinical staff to identify and refer to relevant community resources to address patients' social barriers; implementing a champion within practice to integrate referral into usual care; use of electronic health records to prompt provider referral and share information between provider and the community; and developing a screening process and promotional material to prompt referral.

The ARC project will build on this work by focussing on improving access to community resources in patients' language of choice and emphasizing access to French-language resources for Francophones in Ontario. That component will be established in the Champlain Local Health Integration Network (LHIN). The proposed work will build on team members' experience, the foundational work and existing partnerships established by Dr. Dahrouge and her team.

Hypothesis leading to the present study

Based on the work done to date, we have determined it is warranted to a study an intervention to optimize equitable access to community resources for Ontarians based on the following activities:

1. Improving referrals to community resources by

   * Raising population and providers' awareness of community resources and the existing navigation tools that can help identify where the services are delivered.
   * Engaging the participation of members of the vulnerable communities, including Francophones living in minority situations, and care delivery personnel in our work.
   * Training staff in primary care practices on the use of the electronic and telephone navigation tools
   * Supporting practices to adopt processes that will allow them to incorporate community services into the basket of services they already coordinate (e.g. specialty care)
2. Improving the continuity of care across the two sectors (primary care and community services) by

   - Establishing communication and coordination processes between the primary care practices and the patient navigator.
3. Supporting individuals with social complexities to overcome barriers to adequately access by

   * Increasing awareness of the resources within communities at higher risk of poor access (including Francophones living in minority situations)
   * Providing support to these individuals in the form of a "Navigator" to assist them in overcoming barriers to access.

ELIGIBILITY:
Inclusion Criteria:

Primary care practices:

Four to six practices will be recruited to participate in this feasibility study.The eligibility criteria are:

* A primary care practice, other than Community Health Centre, is eligible regardless of the type of model to which it belongs (Solo, groupe based (Family Health Groups, Family Health Networks, Family Health Organizations), and interprofessional teambased (Family Health Teams)
* Having at least one primary care provider agreeing to participate in the study Primary care members Primary care members working in a participating practice will be invited to participate in the study.

Members are eligible if they can refer practice patients to community resources or staff members who can be involved in the referral process (including nurses, allied health professionals (e.g. social workers), and front desk staff).

For the purpose of simplicity all these are referred to as primary care providers in the document

Patients:

Primary care patients participating in the intervention are eligible to participate if the following criteria are met:

* Patient identifies a primary care provider participating in the study as their main primary care provider
* Has received a recommendation for a community resource from their primary care provider during a primary care encounter
* Is able to communicate in English or French, or is willing to be served via a cultural interpreter.

Patient agrees to participate in the study (18 years of age or older), or has parental/guardian proxy consent to participate in the study (minor patients, patients with cognitive deficits rendering them unable to provide consent, or patients unable to adequately understand French or English to provide informed consent and unable/unwilling to use the services of a translator).

Exclusion Criteria:

* There are no exclusion criteria for primary care providers.

Primary care practices:

* A Community Health Centre
* Practices that are not part of a reform model

Patients:

• Patient has cognitive limitation that would not permit them to give consent and does not have a family member/guardian who can provide proxy consent There are no age, language or other requirements for patient eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Active Patient Utilization | 12 month
  Number of community resources utilized amongst patients who could have referred during that 12 months period. Therefore, it is the number of community resources utilized by practice patients that have had a visit to the practice during the 12 months recruitment period in the practice Total # of services utilized

SECONDARY OUTCOMES:
Referrals | 12 month
  The number of patients referred will be determined based on the referral forms completed. Primary care providers are asked to complete a referral form for all referrals they make to a community resource. The primary care provider then explains that a study is being done, and asks the patient for verbal consent to be contacted by the study team. All referrals having been made, regardless of the patient's interest in participating in the study will be captured. (Referral forms completed for all patients referred to a community resource will be collected by the research team. Patients' name and contact information will appear on referral forms ONLY for patients that consented to this information being provided to the research team).
First Contact Access | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section A in patient survey
Needs/Difficulties/Use of healthcare | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section B in patient survey
Health care experienced | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section C in patient survey
Quality of Life VR12 | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section E in patient survey
Self Efficacy | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section F in patient survey
Engagement with primary medical care and appropriateness of care | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section G in patient survey
Ability to engage | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section H in patient survey
Health Action Process Approach | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section O in patient survey
Patient Activation Measure | baseline (i.e. the time of referrals (Pre-intervention) as well six months later, at the end of the patient six months intervention period .
  Section P in patient survey

CONTACTS AND LOCATIONS:
Locations (1):
- West Ottawa Nepean Family Health Organization, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dahrouge S, Gauthier A, Chiocchio F, Presseau J, Kendall C, Lemonde M, Chomienne MH, Perna A, Toal-Sullivan D, Devlin RA, Timony P, Prud'homme D. Access to Resources in the Community Through Navigation: Protocol for a Mixed-Methods Feasibility Study. JMIR Res Protoc. 2019 Jan 24;8(1):e11022. doi: 10.2196/11022. PMID 30679151